CLINICAL TRIAL: NCT00301015
Title: Rapid Diagnostic Testing and Artemisinin-Based Combination Therapy for Uncomplicated Malaria by Community Health Workers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Collaborators: Muhimbili University of Health and Allied Sciences (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: RapAct 28-02-2006
Record Dates: First submitted 2006-03-08; First posted 2006-03-10 (Estimated); Last update posted 2007-11-01 (Estimated); Status verified 2007-10

CONDITIONS: Uncomplicated Plasmodium Falciparum Malaria
MeSH Terms: interventions — Rapid Diagnostic Tests

ARMS (2):
- 1 (Experimental): Malaria diagnosis aided with rapid diagnostic test
  Interventions: Device: Rapid diagnostic test for malaria
- 2 (Active Comparator): Malaria diagnosis based on clinical judgement only
  Interventions: Device: Rapid diagnostic test for malaria

INTERVENTIONS:
Device: Rapid diagnostic test for malaria — We used Paracheck Pf® (Orchid Biomedical Systems, India) as rapid diagnostic test in this trial

SUMMARY:
The purpose of this study is to evaluate the efficiency of a rapid diagnostic test (Paracheck Pf) for the diagnosis of uncomplicated Plasmodium falciparum malaria by community health workers at village level in Tanzania and how the use of rapid diagnostic test may influence prescription of antimalarial drugs.

The hypothesis is that rapid diagnostic tests used by community health workers will reduce the use of antimalarial drugs (Coartem; Novartis) by 30% without affecting the health outcome.

ELIGIBILITY:
Inclusion Criteria:

* Fever
* Informed consent

Exclusion Criteria:

* Severe clinical manifestations, which require immediate referral
* Pregnancy
* Previous enrollment in the study within the last 28 days

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3005 (Actual)
Dates: Start 2006-03; Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Number of patients with fever prescribed artemether-lumefantrine for the treatment of malaria in respective study groups | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Anders Björkman, MD, PhD, Study Director — Dept of Medicine, Karolinska University Hospital, 171 76 Stockholm, Sweden
Locations (1):
- Villages, Kibaha, Kibaha District, Tanzania

REFERENCES:
- [Derived] Mubi M, Janson A, Warsame M, Martensson A, Kallander K, Petzold MG, Ngasala B, Maganga G, Gustafsson LL, Massele A, Tomson G, Premji Z, Bjorkman A. Malaria rapid testing by community health workers is effective and safe for targeting malaria treatment: randomised cross-over trial in Tanzania. PLoS One. 2011;6(7):e19753. doi: 10.1371/journal.pone.0019753. Epub 2011 Jul 5. PMID 21750697